CLINICAL TRIAL: NCT07140315
Title: An Open-label, Single-center Clinical Trial of [18F]DK222 PET/CT for Imaging of Patients With Non-Small-Cell Lung Cancer (NSCLC) and Urothelial Cancer Who Are Eligible for Treatment With Anti-PD(L)-1
Brief Title: DK222 Study at Hopkins
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J24119; IRB00462780 (Other: Johns Hopkins IRB)
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer; Urothelial Cancer
Keywords: PD-L1; PD-1; PET; Imaging; MSCLC; UC; bladder cancer; lung cancer; radiotracer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]DK222 radiotracer (Experimental): The study is an open label, single-arm study designed to evaluate the safety and diagnostic performance of [18F]DK222 radiotracer in NSCLC and UC participants. Participants will undergo a PET-CT scan after [18F]DK222 is injected into the participant's vein an intravenous line. This is the imaging procedure to assess where [18F]DK222 has accumulated in the body.
  Interventions: Drug: [18F]DK222 radiotracer

INTERVENTIONS:
Drug: [18F]DK222 radiotracer — [18F]DK222 is an investigational radiotracer used detect non-small cell lung cancer (NSCLC) or Urothelial Cancer (UC) tissue in the body when used with positron emission tomography/computed tomography. Participants will undergo a PET-CT scan after [18F]DK222 is injected into the participant's vein an intravenous line.

SUMMARY:
This Phase 1 clinical trial will test a new drug called [18F]DK222 in people with cancer. The goal is to see if the drug is safe, how it spreads through the body, how long it stays in the body, and how much radiation it gives off. [18F]DK222 is designed to attach strongly and specifically to a protein called PD-L1, which helps cancer hide from the immune system.

This is a first in human study to collect preliminary safety and toxicity data of [18F]DK222.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must sign informed consent prior to inclusion in this trial.
* Subjects must be ≥18 years of age and competent to give informed consent.
* Subjects must be diagnosed with histologically confirmed NSCLC or UC and eligible for anti-PD(L)-1 therapy.
* PD-L1 immunohistochemistry result using a Clinical Laboratory Improvement Amendments (CLIA) assay must be available or if not available then sufficient tissue must be available to perform PD-L1 testing.
* Subjects must score at least 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Subjects must have adequate organ function as defined by the following laboratory values (determined within 28 days prior to randomization/registration) or as deemed not clinically significant by physician on record:

  * White blood cells (WBC) ≥ 2000 /μL
  * Absolute neutrophil count (ANC) ≥ 1500 /μL
  * Platelets ≥ 100 x103 /μL
  * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L
  * Serum creatinine ≤ 1.5 times upper limit of normal (ULN) or creatinine clearance greater than or equal to 60 ml/min (using the Cockcroft-Gault formula)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times ULN
  * Bilirubin ≤ 1.5 times ULN (Except patients with the Gilbert Syndrome, for whom a maximum of ≤ 3.0 mg/dL is acceptable)
* Women of childbearing potential (WOCBP) should have a negative serum pregnancy test within 24 hours prior to receiving the first administration [18F]DK222. Women with non-childbearing potential may be included if either surgically sterile or have been postmenopausal for ≥ 1 year.
* WOCBP and men who are sexually active with WOCBP must agree to use appropriate method(s) of contraception.

Exclusion Criteria:

* Prior treatment, in either de novo disease or during this recurrence, with an anti-PD-L1 or anti-PD-L2 antibody. A minimum of 4 month washout period is required for patients treated with anti-PD-L1 or anti-PD-L2 therapy. Patients with disease that was previously treated with anti-PD-1, anti-PD-L1, anti-PD-L2 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, but now have a new recurrence, would be eligible.
* Subjects who have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 Grade 1 or better from the adverse events due to previous cancer therapy.
* Treatment with corticosteroids in an increasing dosage in the 7 days prior to the first administration of anti-PD1. (A stable or decreasing dosage of ≤ 10 mg dexamethasone or equivalent is allowed. In addition, inhaled or topical steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease.)
* A severe hypersensitivity reaction to prior treatment with a monoclonal antibody, or known hypersensitivity to study drugs components.
* Any serious or uncontrolled medical disorder or active infection that, in the opinion of the investigator, may increase the risk associated with study participation, study drug administration, or would impair the ability of the patients to receive protocol therapy.
* Women of childbearing potential with a positive serum or urine pregnancy test (minimum sensitivity 10 IU/L or equivalent units of HCG) within 24 hours prior to the start of imaging.
* Breastfeeding women.
* Inability to comply with other requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety of [18F]DK222 as assessed by number of grade 3-5 adverse events | Once up to 10 days post radiotracer injection
  Any grade 3-5 toxicity attributed to [¹⁸F]DK222 administration will be considered as not meeting the safety endpoint. All adverse events (AEs) will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Tolerability of [18F]DK222 as assessed by number of grade 3-5 adverse events | Once up to 10 days post radiotracer injection
  . Any grade 3-5 toxicity attributed to [¹⁸F]DK222 administration will be considered as not meeting the tolerability endpoint. All adverse events (AEs) will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Ali Mosallaie, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States